CLINICAL TRIAL: NCT05756660
Title: Cisplatin and Sodium Thiosulfate Otoprotection With or Without SAHA/Vorinostat Histone Deacetylase Inhibition for Relapsed/Refractory Hepatoblastoma and Other Embryonal Tumors
Brief Title: Sodium Thiosulfate Otoprotection During Salvage Cisplatin Therapy
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This study will be closing at CCHMC and may be transferred to a principal investigator at another insitutiton.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSS-JG-2201
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Ototoxicity, Drug-Induced
Keywords: Cisplatin; Sodium Thiosulfate; Relapsed/Refractory Hepatoblastoma; PedMark; Embryonal Tumor
MeSH Terms: conditions — Ototoxicity; Hepatoblastoma; Neoplasms, Germ Cell and Embryonal | interventions — sodium thiosulfate; Cisplatin; Vorinostat

STUDY DESIGN:
Intervention Model Description: Three strata are identified for this study:
  Stratum 1: Cisplatin sensitive/no progression on cisplatin (when given at first diagnosis): Regimen Cisplatin/STS (CS)
  Stratum 2A: Cisplatin resistant or progressed on cisplatin after initial response (when given at first diagnosis): Regimen Cisplatin/STS/SAHA (CSS)
  Stratum 2B: Wilms tumor, Germ Cell tumor, Neuroblastoma: Regimen CSS
  Within each of the 3 eligible strata, patients will be enrolled and directly assigned to their respective protocol therapy, yielding 3 independent single-arm cohorts. Patients will receive protocol therapy for up to 6 3-week cycles before moving to follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Stratum 1- Regimen CS (Experimental): Cisplatin sensitive/no progression on cisplatin (when given at first diagnosis)
  Interventions: Drug: Sodium Thiosulfate
- Stratum 2A- Regimen CSS (Experimental): Cisplatin resistant or progressed on cisplatin after initial response (when given at first diagnosis)
  Interventions: Drug: Sodium Thiosulfate
- Stratum 2B- Regimen CSS (Experimental): Wilms tumor, GCT, Neuroblastoma
  Interventions: Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Sodium Thiosulfate — This goal of this study is to evaluate the efficacy of the proposed regimens in patients with relapsed/refractory platinum pre-treated patients with Hepatoblastoma, Wilms tumor, Germ Cell Tumor (GCT), and Neuroblastoma. The patients' initial cisplatin response (hepatoblastoma) and diagnosis will determine their treatment regimen on this study.
  Other Names: Cisplatin; Vorinostat/ SAHA

SUMMARY:
This study will attempt to demonstrate the efficacy of Sodium Thiosulfate (STS) in preventing hearing loss in patients re-treated with cisplatin-based therapy according to regimens Cisplatin and STS (regimen CS) and Cisplatin, STS and Vorinostat/SAHA (regimen CSS).

DETAILED DESCRIPTION:
This trial will assess the effect of STS in preventing subsequent hearing loss when patients are re-challenged with cisplatin therapy at relapse/progression, as well as the efficacy of cisplatin/STS or cisplatin/STS/SAHA for patients with relapsed hepatoblastoma, Wilms, Germ Cell Tumor (GCT) and Neuroblastoma stratified by initial cisplatin sensitivity. Important pharmacokinetic measurements focused on cisplatin and STS in children, with varying degrees of renal function, will be assessed. Such pharmacokinetic data will fill a current gap in our clinical knowledge base and enable safer use of such agents for all children with such cancers, regardless of kidney function, in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 1 month and ≤ 39 years old at study enrollment
* Histologically proven, at time of diagnosis or relapse:

  1. Stratum 1: Arm CS (Cisplatin/STS): Previously chemosensitive to cisplatin defined as an AFP drop of 1 log (90%) and/or an objective tumor response of 30% or greater on imaging while receiving cisplatin.
  2. Stratum 2A: Cisplatin/STS/SAHA (CSS): Previously chemosensitive but with noted subsequent progression on cisplatin or initially chemoresistant to cisplatin (all other hepatoblastoma patients). Resistance to cisplatin is defined as rising alpha-fetoprotein (AFP) x 2 consecutive measurements or imaging progression including growth of known lesions or new lesions while patient is receiving a cycle of chemotherapy containing cisplatin or relapse noted within 3 months of last cisplatin administration.
  3. Stratum 2B: CSS: Relapsed/refractory Wilms tumor, Germ Cell Tumor, or Neuroblastoma
* Patients must have a life expectancy of ≥ 8 weeks.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study:

  1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study. Previous SAHA administration is permitted. Tacrolimus and Sirolimus with levels <= 10 ng/ml are not considered myelosuppressive.
  2. Immunotherapy: Must not have received within 2 weeks of entry onto this study.
  3. Radiation therapy (RT): greater than or equal to 2 weeks for local palliative RT (small port); greater than or equal to 6 months must have elapsed if prior craniospinal RT or if greater than or equal to 50% radiation of pelvis
* Patients may not be enrolled on another clinical trial or receiving any other investigational therapies (within 2 weeks prior to study enrollment).
* Organ Function Requirements

  1. Adequate Bone Marrow Function Defined as:

     1. Peripheral absolute neutrophil count (ANC) greater than or equal to 750/uL
     2. Platelet count greater than or equal to 75,000/uL (transfusion independent defined as no platelet transfusions within 7 days)
     3. Hemoglobin greater than or equal to 8.0 g/dL (may receive red blood cell transfusions)
  2. Adequate Liver Function Defined As:

     1. Total OR direct bilirubin less than or equal to 1.5 x upper limit of normal (ULN) for age, and
     2. Aspartate aminotransferase (AST) or Alanine transaminase (ALT) < 10x ULN
  3. Adequate Renal Function Defined As:

     1. Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 30 mL/min/1.73 m2
* Baseline Audiology Requirements:

  1. Subjects must have a successful audiology examination prior to enrollment. Patients may have Boston grade III or IV hearing loss and still be eligible to enroll as long as they did not receive 3 or more cycles of cisplatin during upfront therapy WITH sodium thiosulfate. There is no specific baseline hearing level/grade requirement beyond that to be eligible, but the baseline level of hearing must be clearly established and recorded

Exclusion Criteria:

* Patients with any uncontrolled, intercurrent illness including, but not limited to, uncontrolled infection
* Patients with symptomatic congestive heart failure (defined as Grade 2 or higher heart failure per CTCAE version 5.0)
* Patients with Renal Tubular Acidosis (RTA) as evidenced by serum bicarbonate < 16 mmol/L and serum phosphate ≤ 2 mg/dL (or < 0.8 mmol/L) without supplementation. Patients requiring electrolyte supplementation for RTA will be permitted if bicarbonate ≥16 mmol/L and phosphate > 2mg/dL after at least 7 days of stable supplementation regimen
* Pregnancy and Breastfeeding:

  1. Female patients who are pregnant or breast-feeding will not be entered in the study. A negative pregnancy test within 72 hours of starting therapy is required for female patients of childbearing potential
  2. Lactating females who plan to breastfeed their infants.
  3. Sexually active patients of reproductive potential must agree to use an effective contraceptive method for the duration of their study participation
* Patients on tacrolimus and/or sirolimus with levels of either targeted > 10 ng/mL
* Known allergy to any component of CS or CSS therapy, as indicated

Ages: 1 Month to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of hearing loss | Through study completion up to 5 years
  To demonstrate the efficacy of Sodium Thiosulfate (STS) in preventing hearing loss in patients re-treated with cisplatin-based therapy according to regimens Cisplatin/STS (CS) and Cisplatin/STS/SAHA (CSS)

SECONDARY OUTCOMES:
Prevention of hearing loss and tumor reduction | Through study completion up to 5 years
  Number of patients with minimal hearing loss as measure by audiogram evaluations. Number of patients with positive tumor response as measured by Response Evaluation Criteria in Solid Tumors (RECIST).
Number of Participants with Treatment-Related Adverse Events | Through study completion up to 5 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Stratum 1 efficacy | Through study completion up to 5 years
  Arm A/CS: To describe the clinical efficacy of CS, as defined by objective response, in patients with relapsed/refractory Hepatoblastoma that was initially sensitive to cisplatin and without progression on cisplatin
Stratum 2 efficacy | Through study completion up to 5 years
  To define the clinical efficacy of CSS, as defined by objective response, in patients with initial cisplatin refractory Hepatoblastoma or in patients who progress on cisplatin
Maximum Plasma Concentration [Cmax] | Through study completion up to 5 years
  To investigate the concentration of cisplatin in patients with varying degrees of renal dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Somers, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cincinnati Children's Hospital Medical Center home page — http://www.cincinnatichildrens.org/service/c/cancer-blood